CLINICAL TRIAL: NCT01153074
Title: Bronchoscopic Closure of Bronchopleural Fistulas With Occlutech Figulla ASD N Occluder Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: InCor Heart Institute (Other); Occlutech International AB (Industry)
Responsible Party: Principal Investigator, Miguel L. Tedde, MD, PhD, University of Sao Paulo
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: USP01089/09-TBF
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Bronchopleural Fistula
Keywords: Bronchopleural fistula; Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Occluder (Experimental): The patients with bronchopleural fistulas treated with bronchoscopic deployment of the cardiac septal defects occluder.
  Interventions: Device: Closure of bronchopleural fistula with Occlutech Figulla

INTERVENTIONS:
Device: Closure of bronchopleural fistula with Occlutech Figulla — Patients with bronchopleural fistulas will be submitted to a bronchoscopic procedure to deploy the cardiac septal defect occluder in the fistula traject.
  Other Names: Bronchoscopic bronchopleural fistula closure with occluders

SUMMARY:
The purpose of this study is to evaluate the feasibility of closing bronchopleural fistulas with devices originally developed for correction of cardiac septal defects deployed through bronchoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 14 years old
* Bronchopleural fistulas

Exclusion Criteria:

* Clinical conditions increasing surgical risk (hemodynamic instability, respiratory distress)
* Immunosuppressed patients
* Acute intense inflammatory process in fistula edge
* Suppurative pleural cavity infection

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-06; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Closure of tracheobronchial fistulas with the Occlutech Figulla ASD N occluder | 1 year
  The closure of the fistulas will be bronchoscopically observed at regular intervals: one week, three weeks, two months and six months.
  At the third months post intervention, a thorax CT scan will ascertain the correct position and stability of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel L. Tedde, MD, PhD, Principal Investigator — Heart Institute (InCor) HC of the Sao Paulo University School
Locations (2):
- Brazil (2):
  - Heart Institute (InCor) Hospital das Clinicas, Faculdade de Medicina, Universidade de Sao Paulo, São Paulo
  - Hospital das Clinicas, Faculdade de Medicina, Universidade de Sao Paulo, São Paulo

REFERENCES:
- [Result] Tedde ML, Scordamaglio PR, Rodrigues A, Minamoto H, Alfinito FS. Minimally invasive closure of bronchopleural fistulas. Chest. 2011 Sep;140(3):826. doi: 10.1378/chest.11-0719. No abstract available. PMID 21896530
- [Result] Tedde ML, Minamoto H, Scordamaglio PR, Rodrigues A, Moura EG, Pedra CA. Broncoscopic closure of tracheoesophageal fistulas. Ann Thorac Surg. 2011 Apr;91(4):1311. doi: 10.1016/j.athoracsur.2010.09.015. No abstract available. PMID 21440188
- [Result] Scordamaglio PR, Tedde ML, Minamoto H, Pedra CA, Jatene FB. Endoscopic treatment of tracheobronchial tree fistulas using atrial septal defect occluders: preliminary results. J Bras Pneumol. 2009 Nov;35(11):1156-60. doi: 10.1590/s1806-37132009001100015. English, Portuguese. PMID 20011853
- [Result] Scordamaglio PR, Tedde ML, Minamoto H, Assad RS, Fernandes PMP. Can total bronchopleural fistulas from complete stump dehiscence be endoscopically treated? Eur J Cardiothorac Surg. 2017 Apr 1;51(4):702-708. doi: 10.1093/ejcts/ezw377. PMID 28082466